CLINICAL TRIAL: NCT07152561
Title: Effect of Two Different Luting Cements on Clinical Outcomes of Pediatric Zirconia Crowns: A Randomized Controlled Trial
Brief Title: Different Luting Cements for Pediatric Zirconia Crowns
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rasha Mohamed Hatem Hanafy, Associate Professor of Pediatric Dentistry and Dental Public Health, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pediatric Zirconia Crowns
Record Dates: First submitted 2025-08-26; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Dental Caries in Children
MeSH Terms: interventions — Resin Cements

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Zirconia crown cemented with Predicta® Bioactive Cement
  Interventions: Drug: Zirconia crown cemented with Predicta® Bioactive Cement
- Arm 2 (Active Comparator): Zirconia crown cemented with resin-cement
  Interventions: Drug: Zirconia crown cemented with resin-cement

INTERVENTIONS:
Drug: Zirconia crown cemented with Predicta® Bioactive Cement — • For the bioactive cement group (Predicta® Bioactive Cement), the prepared tooth will be dried using compressed air but not desiccated. Cement will be dispensed through the auto-mixtip directly into the crown, and the crown will be properly positioned over the tooth; cement will be allowed to self-set for 20 seconds while maintaining gentle pressure on the crown. Buccal and lingual margins will be flash-cured for 10 seconds each using a light-curing unit to immediately cure the excess cement for easier removal, and buccal and lingual surfaces will then be light-cured for an extra 10 seconds each.
  Arms: Arm 1
Drug: Zirconia crown cemented with resin-cement — • For the resin-cement group, the tooth will be dried with compressed air but not desiccated. The sealant will be applied with the syringe; then, the crown will be appropriately positioned over the tooth, and cement will be allowed to self-set for 2 minutes and cured while maintaining gentle pressure on the crown. Excess cement will be removed before the cement is completely set.
  Arms: Arm 2

SUMMARY:
The study aims to compare the efficacy of using bioactive cement versus resin-cement for cementation of anterior pediatric zirconia crowns.

DETAILED DESCRIPTION:
* For the bioactive cement group (Predicta® Bioactive Cement), the prepared tooth will be dried using compressed air but not desiccated. Cement will be dispensed through the auto-mixtip directly into the crown, and the crown will be properly positioned over the tooth; cement will be allowed to self-set for 20 seconds while maintaining gentle pressure on the crown. Buccal and lingual margins will be flash-cured for 10 seconds each using a light-curing unit to immediately cure the excess cement for easier removal, and buccal and lingual surfaces will then be light-cured for an extra 10 seconds each.
* For the resin-cement group, the tooth will be dried with compressed air but not desiccated. The sealant will be applied with the syringe; then, the crown will be appropriately positioned over the tooth, and cement will be allowed to self-set for 2 minutes and cured while maintaining gentle pressure on the crown. Excess cement will be removed before the cement is completely set.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had no history of allergies
* Children who had at least two carious primary incisors.
* Teeth with multi-surface carious lesion.
* Teeth with no percussion or palpation sensitivity
* Teeth with no abscess and/or fistula
* Teeth with no prior pulpal treatment
* Teeth with no mobility or signs of periodontal disease

Exclusion Criteria:

* Children with congenital developmental defects (such as amelogenesis imperfecta and dentinogenesis imperfecta)
* Children with a history of bruxism, trauma or infraocclusion
* Children with a skeletal or dental malocclusion

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-08-28 (Estimated); Primary Completion 2026-08-28 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Retention | 1 week, 1 month, 3 months, 6 months, 9 months, and 12 months
  Retention will be assessed by visual inspection and probe to detect debonded crowns.
Fracture | 1 week, 1 month, 3 months, 6 months, 9 months, and 12 months
  Fractures will be assessed using visual inspection to detect incomplete fracture lines or complete fractures with loss of crown material.

SECONDARY OUTCOMES:
The gingival condition | 1 week, 1 month, 3 months, 6 months, 9 months, and 12 months
  The gingival condition around cemented crowns will be assessed by calculating the gingival index for each crowned tooth.